CLINICAL TRIAL: NCT02520297
Title: A Phase 2, Open-label Pilot Study of TRV130 for the Treatment of Moderate to Severe Acute Pain Associated With Long Bone Fracture
Brief Title: A Pilot Study of TRV130 for the Treatment of Fracture Pain
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Trevena Inc. (Industry)
Collaborators: Kestrel Biologic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP130-2004
Record Dates: First submitted 2015-08-07; First posted 2015-08-11 (Estimated); Results first posted 2020-09-07 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-08

CONDITIONS: Pain
Keywords: Pain; Long bone; Fracture
MeSH Terms: conditions — Pain; Fractures, Bone | interventions — ((3-methoxythiophen-2-yl)methyl)((2-(9-(pyridin-2-yl)-6-oxaspiro(4.5)decan-9-yl)ethyl))amine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TRV130 (Experimental): Drug: TRV130
  Interventions: Drug: TRV130

INTERVENTIONS:
Drug: TRV130 — Drug

SUMMARY:
The primary objective is to evaluate the analgesic efficacy of TRV130 for moderate to severe acute pain in patients presenting to the emergency department (ED) with a suspected/known, unilateral, closed long bone fracture.

DETAILED DESCRIPTION:
This study is designed to evaluate the analgesic efficacy of TRV130 for the treatment of moderate to severe acute pain associated with a long bone fracture in patients presenting to the ED. The safety and tolerability of TRV130 will also be evaluated in this open-label pilot study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years, inclusive
* Has a suspected/known, unilateral, closed fracture of either: radius, ulna (or both) OR tibia, fibula (or both) BUT not fractures in more than 1 extremity
* Able to understand and comply with study procedures and requirements, and provide written informed consent

Exclusion Criteria:

* Significant concomitant head, chest, or abdominal trauma
* Multiple extremity trauma
* Open fracture
* Clinically significant medical condition or history of such condition that may place the patient at an unacceptable risk in the trial, may interfere with the interpretation of efficacy, safety, or tolerability data obtained in the trial, or may interfere with the absorption, distribution, metabolism, or excretion of drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-10-20 (Actual); Primary Completion 2015-10-23 (Actual); Study Completion 2015-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Indiana University, Principal Investigator — Indiana University
Locations (1):
- Trevena, Inc., Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TRV130
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | TRV130
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Achieving Clinical Response, Defined as Achieving a NPRS <= 3, Without Requiring Rescue Pain Medication.
Description: Pain intensity will be evaluated using an 11-point numeric pain rating scale administered over 3 hours
Time Frame: 3-hours
Population: Study terminated early. Primary outcome not measured.
Arm/Group | TRV130
Number analyzed (Participants) | 0

2. Secondary Outcome: Time Weighted Average Change in NPRS
Description: Pain intensity will be evaluated using an 11-point numeric pain rating scale administered over 3 hours
Time Frame: From baseline to 30 minutes, to 1 hour, to 2 hours and to 3 hours
Population: Study terminated early. Secondary outcome not measured.
Arm/Group | TRV130
Number analyzed (Participants) | 0

3. Secondary Outcome: Time to First NPRS <= 3
Description: Pain intensity will be evaluated using an 11-point numeric pain rating scale administered over 3 hours
Time Frame: 3-hours
Population: Study terminated early. Secondary outcome not measured.
Arm/Group | TRV130
Number analyzed (Participants) | 0

4. Secondary Outcome: Safety Assessments
Description: Safety assessments include adverse events, vital sign measurements, physical examination findings, and clinical laboratory assessments.
Time Frame: 3-hours
Population: Study terminated early. Secondary outcome not measured.
Arm/Group | TRV130
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | TRV130
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
Study terminated early due to lack of enrollment. Analyses for the primary and secondary outcomes were not completed. No mortalities, serious adverse events, or adverse events were reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other